CLINICAL TRIAL: NCT06989866
Title: Opiate-sparing Post-operative Pain Control in Septorhinoplasty: A Prospective Randomized, Double Blind Clinical Trial
Brief Title: RCT to Test Regional Anesthesia Effect on Decreased Opiate Use
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCP.2024.0031
Record Dates: First submitted 2025-04-10; First posted 2025-05-25 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Experimental): Application of regional block to the nose with Exparel
  Interventions: Drug: Bupivacaine
- Saline (Placebo Comparator): Application of injectable saline to the nose
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Bupivacaine — Bupivicaine injection post operatively
  Arms: Exparel
Drug: Saline (NaCl 0,9 %) (placebo) — Saline injected to control group
  Arms: Saline

SUMMARY:
Examining use of strong pain medication with the use of perioperative anesthetic medications vs no use of the same perioperative medication

DETAILED DESCRIPTION:
Control group:

1. At the end of the Septorhinoplasty while the patient is still under general anesthesia, an associate investigator assisting in the case will administer normal saline to V2 (maxillary branch of the trigeminal nerve superiorly), nasal dorsum, and infraorbital foramen on each side. The total volume will consist of up to 10ml of normal saline. These injections are not standard of care but are performed for research purposes. The injections will be performed under the direct supervision of the staff surgeon, a board certified otolaryngologist. Each AI has performed injections of this nature (method and location) before - not with Exparel but the method and location are the same.
2. Following surgery, the subject will receive handouts including patient informational sheet regarding appropriate use of opioid medications, scheduling acetaminophen and ibuprofen, and a tracking sheet or medication usage. The tracking sheet is provided for study purposes, whereas all other materials are per the standard of care.
3. Oral medications will be prescribed by resident physician per the standard of care guidelines.
4. Subjects will be counseled on return precautions and will be given contact information for routine and emergency visits (standard of care).
5. Patients will be instructed to return in one week for removal of the intraoperative splint placement (standard of care) and bring the tracking sheets and medications with them (research purposes only).

Treatment group:

1. At the end of the Septorhinoplasty while the patient is still under general anesthesia, an associate investigator assisting in the case will administer liposomal bupivacaine (Exparel) to V2 (maxillary branch of the trigeminal nerve superiorly), nasal dorsum, and infraorbital foramen on each side. The total volume will be the same as the control group: up to 10mL. These injections are not standard of care but are performed for research purposes. The injections will be performed under the direct supervision of the staff surgeon, a board-certified otolaryngologist. Each AI has performed injections of this nature (method and location) before - not with Exparel but the method and location are the same.
2. Following surgery, the patient will receive handouts including patient informational sheet regarding appropriate use of opioid medications, scheduling acetaminophen and ibuprofen, and a tracking sheet for medication usage. The tracking sheet is provided for study purposes, whereas all other materials are per the standard of care.
3. Medications will be prescribed by resident physician per the standard of care guidelines.
4. Patients will be counseled on return precautions and will be given contact information for routine and emergency visits (standard of care).
5. Patients will be informed to return in one week for removal of the intraoperative splint placement (standard of care) and bring the tracking sheets and pill bottles with them (research purposes only).

Both Control and Treatment groups:

Per NMCP policy, a teal-colored wrist band will be placed on all study participants following surgery indicating that Exparel was administered, even for those that did not receive Exparel. Subjects will be instructed not to remove the band for at least 96 hours (4 days) following surgery. All participants receive this band to maintain the blinding of the study. Local anesthetics, even topical (applied to the skin), should generally be avoided within 96 hours (4 days) of surgery. Should the subject seek emergency care at an outside facility in the 7 days following surgery, they will be instructed to inform providers that they are participating in a research study and may have received Exparel. If the provider has any questions or concerns, the subject will provide them with the ENT Duty contact information. The need for emergency care for post-septorhinoplasty patients is rare, and in most cases they will return to NMCP, but in the event they do not instructions will be provided to contact the NMCP ENT team. If the provider on duty is not an investigator on the study, they will contact a member of the study team to determine if the subject in question is part of the treatment or control group to help determine their care at the outside facility.

Follow-up:

1. Patients will return for removal of their intranasal splints at approximately one week postop (standard of care).
2. During this encounter medication tracking sheets (DCT 003) will be collected, and a validated pain survey (PROMIS - Patient-Reported Outcome Measurement Information System, DCT 002) will be administered in office for research purposes. The PROMIS questionnaire has been amended to only include the 3 questions needed for this study.
3. Investigators will record the total pills remaining from opioid prescription for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a primary septorhinplasty at NMCP or Langley Air Force Base

Exclusion Criteria:

* History of alcohol abuse/dependence, mental health medications or opiate use disorder. Revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Use of Opiate Pain Medications After Rhinoplasty | 1 week
  How many opiate pills are used after rhinoplasty

SECONDARY OUTCOMES:
PROMIS - Pain Intensity Questionnaire | 1 week
  Recording pain scale after surgery for 1 week, A score of 1 equals no pain/good outcome, score of 5 equals severe pain/worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tokunbo I Ayeni, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: No